CLINICAL TRIAL: NCT01593917
Title: Long Term Follow Up Study of the St. Jude Medical Trifecta™ Valve
Brief Title: Trifecta™ Long Term Follow-Up (LTFU) Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 1104
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Regurgitation; Aortic Valve Stenosis; Aortic Valve Incompetence
Keywords: Aortic valve; Heart valve; Tissue valve; Bioprosthesis
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects previously implanted with a Trifecta™ valve in the Trifecta™ IDE Study: Subjects enrolled in this clinical study were implanted with the Trifecta™ aortic bioprosthetic valve during 2007, 2008 and 2009 as part of the Trifecta™ IDE Study conducted to obtain FDA approval.
  Interventions: Device: Trifecta™ Valve

INTERVENTIONS:
Device: Trifecta™ Valve — Aortic valve replacement with the Trifecta™ aortic bioprosthesis.

SUMMARY:
The Trifecta™ LTFU Study is a single-arm, multi-center, prospective, non-randomized, post-market study conducted in the United States and Canada to collect long-term safety and effectiveness data through 10 years after implant of the Trifecta™ aortic bioprosthetic valve. The Trifecta™ is a tri-leaflet stented pericardial valve designed for supraannular placement in the aortic position. The Trifecta™ LTFU Study is an extension of the Trifecta™ Investigational Device Exemption (IDE) Study (NCT00475709) conducted to support United States Food and Drug Administration (FDA) approval of the Trifecta™ valve. All Trifecta™ LTFU Study subjects received Trifecta™ valve implants during participation in the Trifecta™ IDE study and subsequently consented to extended annual follow-up through 10 years under the Trifecta™ LTFU protocol.

DETAILED DESCRIPTION:
This clinical study was designed as an extension of the Trifecta™ IDE Study supporting FDA approval of the Trifecta™ valve. A total of 11 Trifecta™ IDE Study investigational sites in the United States (n=9) and Canada (n=2) participated in the Trifecta™ LTFU Study. Study enrollment included 329 subjects implanted from 2007 through 2009 at these 11 sites during the IDE Study who consented to participate in continued annual follow-up through 10 years post-implant. Of these 329 subjects, 140 also participated in the FDA-mandated Trifecta™ Post-Approval Study (PAS, NCT01514162) prior to consenting to additional annual follow-up under the Trifecta™ LTFU protocol. The remaining 189 subjects entered the Trifecta™ LTFU Study directly from the Trifecta™ IDE Study.

The Trifecta™ LTFU Study database subsumes all data collected in the 329 participants under the Trifecta™ IDE and Trifecta™ PAS protocols and extends these data through 10 years from each subject's original date of implant in the Trifecta™ IDE Study. The Trifecta™ LTFU Study data thus encompass 10 years of continuous annual post-implant follow-up in the 329 participants as well as their pre-implant Baseline Visit data. Data collected includes adverse events, assessments of heart failure symptoms by New York Heart Association (NYHA) functional classification, and echocardiographic assessments of Trifecta™ valve function.

ELIGIBILITY:
Inclusion Criteria:

1. Patient currently has a Trifecta™ aortic valve that was implanted at one of the U.S. or Canadian investigational sites during the Trifecta™ IDE study.
2. Patient met eligibility criteria prior to enrollment in the Trifecta™ IDE study.
3. Patient agrees to complete all required follow-up visits.
4. Patient provided written informed consent prior to any study related procedure, as approved by the governing Institutional Review Board (IRB) or the Ethics Committee (EC) of the investigational site.

Exclusion Criteria:

1. Patient is currently participating or planning to participate in any other study unless approved by the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously implanted with a Trifecta prosthetic valve
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart
Locations (11):
- United States (9):
  - USC University Hospital, Los Angeles, California
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mission Health & Hospitals, Asheville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Main Line Health Center/Lankenau Hospital, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Salt Lake Cardiovascular and Thoracic Surgery, Salt Lake City, Utah
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Institut de Cardiologie de Quebec (HÃ´pital Laval), Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bavaria JE, Desai ND, Cheung A, Petracek MR, Groh MA, Borger MA, Schaff HV. The St Jude Medical Trifecta aortic pericardial valve: results from a global, multicenter, prospective clinical study. J Thorac Cardiovasc Surg. 2014 Feb;147(2):590-7. doi: 10.1016/j.jtcvs.2012.12.087. Epub 2013 Mar 7. PMID 23477687
- [Background] Goldman S, Cheung A, Bavaria JE, Petracek MR, Groh MA, Schaff HV. Midterm, multicenter clinical and hemodynamic results for the Trifecta aortic pericardial valve. J Thorac Cardiovasc Surg. 2017 Mar;153(3):561-569.e2. doi: 10.1016/j.jtcvs.2016.09.089. Epub 2016 Nov 18. PMID 27964975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 329 subjects were enrolled into the Trifecta™ Long Term Follow-Up (LTFU) Study at 11 sites in the United States and Canada. All 329 subjects had received Trifecta™ implants in 2007, 2008 and 2009 during their participation in the Trifecta™ Investigational Device Exemption Study (IDE) Study (NCT00475709). Trifecta™ LTFU study enrollments occurred between 02 July, 2012 and 27 March, 2017. The final 10-years post-Trifecta™-implant follow-up visit was completed on 26 September, 2019.
Pre-assignment Details: The 329 subjects participated in the pre-market Trifecta™ IDE Study used to obtain Food and Drug Administration (FDA) approval. Thereafter, they consented to extended follow-up in the Trifecta™ LTFU Study. Additionally, 140 of the 329 participated in the FDA-required Trifecta™ Post-Approval Study (PAS, NCT01514162) before entering the LTFU Study. Trifecta™ LTFU data subsume the 329 subjects' data from the IDE and PAS protocols and extend these data through 10-years from Trifecta™ implant.
Groups:
- Subjects Previously Implanted With a Trifecta™ Valve: Subjects enrolled in this clinical study received the Trifecta™ valve during the Trifecta™ IDE Study conducted to obtain FDA approval.
Period: Overall Study
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Started | 329
Completed | 159
Not Completed | 170
Not completed — Death | 67
Not completed — Valve-in-valve Transcatheter Aortic Valve Implantation (TAVI) or Surgical Explant | 60
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 12
Not completed — Protocol Violation | 5
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Previously Implanted With a Trifecta™ Valve: Subjects enrolled in this clinical study were implanted with the Trifecta™ valve in 2007, 2008 and 2009 as part of the Trifecta™ IDE Study conducted to obtain FDA approval. Baseline data are from the pre-implant Baseline and Implant Visits in the Trifecta™ IDE Study.
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 224
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 102
  United States | 227
Preoperative New York Heart Association (NYHA) functional classification III or IV [Count of Participants; unit: Participants] — NYHA functional classification is a widely used four class ( I, II, III, and IV) measure of the severity of heart failure symptoms. Class I and II patients experience no or slight limitations on their physical activity. Class III and IV patients experience marked limitations on their physical activity or are unable to perform any physical activity without discomfort.
  Participants | 140
History of Coronary Artery Disease [Count of Participants; unit: Participants] | 180
History of Hypertension [Count of Participants; unit: Participants] | 260
History of Diabetes [Count of Participants; unit: Participants] | 80
History of Smoking [Count of Participants; unit: Participants] | 188
Preoperative Coumarin Derivatives [Count of Participants; unit: Participants] — Coumarin derivatives are anticoagulant medications prescribed to patients at high risk of forming blood clots that can block critical blood vessels. The most widely used coumarin derivative medication is warfarin.
  Participants | 33
Preoperative Aspirin [Count of Participants; unit: Participants] | 228
Preoperative Antiplatelet Medication [Count of Participants; unit: Participants] | 24
Previous Cardiovascular Surgery/Procedure [Count of Participants; unit: Participants] | 85
No Concomitant Procedure [Count of Participants; unit: Participants] | 160
Concomitant Coronary Artery Bypass Grafting (CABG) [Count of Participants; unit: Participants] | 104
Cardiopulmonary Bypass Time (minutes) [Mean (Standard Deviation); unit: minutes] | 103.8 (44.8)
Aortic Cross Clamp Time (minutes) [Mean (Standard Deviation); unit: minutes] | 78.7 (34)
Implanted Valve Size [Count of Participants; unit: Participants]
  19 mm | 22
  21 mm | 78
  23 mm | 113
  25 mm | 86
  27 mm | 24
  29 mm | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Reoperation for Structural Valve Deterioration at 10 Years Post-Implant
Description: Percentage of participants free from surgical explant or valve-in-valve transcatheter aortic valve implantation for treatment of structural deterioration of the Trifecta™ valve through 10 years post-implant. This percentage is estimated from time-to-event data using the Kaplan-Meier estimator. Structural valve deterioration is deterioration intrinsic to the bioprosthetic valve, due to leaflet calcification, leaflet tears, or other causes, that results in prosthetic valve stenosis or regurgitation.
Time Frame: 10 years post-implant
Population: Analysis population includes participants implanted with the Trifecta™ valve in 2007, 2008 and 2009 as part of the Trifecta™ IDE Study who consented to be enrolled in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Subjects Previously Implanted With a Trifecta™ Valve: Subjects enrolled in this clinical study were implanted with the Trifecta™ valve as part of the Trifecta™ IDE Study conducted to obtain FDA approval.
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Percentage of Participants | 75.7 [70.0 to 80.5]

2. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality at 10 Years Post-Implant
Description: Percentage of participants free of death from any cause through 10 years after implant with the Trifecta™ valve, estimated from time-to-event data using the Kaplan-Meier estimator.
Time Frame: 10 years post-implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Percentage of Participants | 77.1 [71.6 to 81.6]

3. Secondary Outcome: Percentage of Participants With Freedom From Valve-Related Mortality at 10 Years Post-Implant
Description: Percentage of participants free from death related to the Trifecta™ valve through 10 years after implant, estimated from time-to-event data using the Kaplan-Meier estimator. Valve-related mortality includes deaths due to any of the following events involving the study valve: structural valvular deterioration, nonstructural valve dysfunction, valve thrombosis, embolism, bleeding events, endocarditis, or reoperation. Sudden, unexplained deaths of participants implanted with the Trifecta™ valve are also counted as valve-related mortality.
Time Frame: 10 years post-implant
Population: Analysis population includes participants implanted with the Trifecta™ valve as part of the Trifecta™ IDE Study who consented to be enrolled in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Percentage of Participants | 98.4 [95.7 to 99.4]

4. Secondary Outcome: Percentage of Participants With Freedom From Structural Valve Deterioration at 10 Years Post-Implant
Description: Percentage of participants free of structural deterioration of the Trifecta valve through 10 years after implant, estimated from time-to-event data using the Kaplan-Meier estimator. Structural valve deterioration is deterioration intrinsic to the bioprosthetic valve, due to leaflet calcification, leaflet tears, or other causes, that results in prosthetic valve stenosis or regurgitation. The presence of structural valve deterioration is determined by direct visualization of the valve at explant or autopsy or by echocardiographic or other cardiac imaging criteria for assessment of valvular stenosis and regurgitation.
Time Frame: 10 years post-implant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Percentage of Participants | 68.4 [62.1 to 73.8]

5. Other Pre Specified Outcome: Number of Late Adverse Events Per 100 Patient-Years of Follow-up
Description: Late adverse events are defined those occurring from 31 days through 10 years post-implant. This outcome measure is calculated by dividing the number of late adverse events of each type by the total number of patient-years of follow-up accumulated from 31 days through 10 years post-implant, expressed in hundreds of years.
Time Frame: 31 days through 10 years post-implant
Population: as for outcome 1
Measure: Number; unit: Number of events per 100 patient-years
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Number of events per 100 patient-years
  All-Cause Mortality | 2.34
  Valve-Related Mortality | 0.17
  Structural Valve Deterioration (SVD) | 2.93
  Reoperation for SVD (surgical explant or transcatheter valve-in-valve implant) | 2.27
  Thromboembolism | 0.52
  Valve Thrombosis | 0.03
  Major Bleeding | 1.05
  Major Paravalvular Leak | 0.00
  Endocarditis | 0.17

6. Other Pre Specified Outcome: Participants' Average Mean Transvalvular Gradient at 10 Years Post-implant by Valve Size
Description: Average of participants' mean aortic transvalvular pressure gradient measured by echocardiography at 10 years post-implant. Averages are reported for each valve size separately. The mean transvalvular pressure gradient is the mean difference in pressure between the inlet side and outlet side of the aortic valve during systole, measured in millimeters of mercury (mmHg).
Time Frame: 10 years post-implant
Population: Analysis population includes participants implanted with the Trifecta™ valve in 2007, 2008 and 2009 as part of the Trifecta™ IDE Study who consented to be enrolled in this study and who have 10-year mean gradient data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 155
mmHg
  19 mm: number analyzed (Participants) | 9
  19 mm | 24.9 (12.4)
  21 mm: number analyzed (Participants) | 39
  21 mm | 17.7 (8.3)
  23 mm: number analyzed (Participants) | 54
  23 mm | 16.0 (9.1)
  25 mm: number analyzed (Participants) | 36
  25 mm | 13.2 (12.4)
  27 mm: number analyzed (Participants) | 13
  27 mm | 8.7 (5.7)
  29 mm: number analyzed (Participants) | 4
  29 mm | 11.0 (3.0)

7. Other Pre Specified Outcome: Participants' Mean Aortic Effective Orifice Area (EOA) Measurement at 10 Years Post-Implant by Valve Size
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve estimated by echocardiography. Mean EOA in square centimeters is reported separately for each valve size.
Time Frame: 10 years post-implant
Population: Analysis population includes participants implanted with the Trifecta™ valve as part of the Trifecta™ IDE Study who consented to be enrolled in this study and who have EOA data available at 10 years post-implant.
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 151
square centimeters
  19 mm: number analyzed (Participants) | 8
  19 mm | 1.0 (0.3)
  21 mm: number analyzed (Participants) | 37
  21 mm | 1.2 (0.3)
  23 mm: number analyzed (Participants) | 53
  23 mm | 1.4 (0.3)
  25 mm: number analyzed (Participants) | 36
  25 mm | 1.7 (0.5)
  27 mm: number analyzed (Participants) | 13
  27 mm | 1.7 (0.4)
  29 mm: number analyzed (Participants) | 4
  29 mm | 1.7 (0.1)

8. Other Pre Specified Outcome: Number of Participants by Aortic Valvular Regurgitation Grade at 10 Years Post-Implant
Description: Regurgitation occurs when the aortic valve does not fully seal, allowing backflow of blood through the closed valve. The amount of aortic regurgitation in this study was graded as none, trivial, mild, moderate or severe by echocardiographic assessment. Moderate or severe aortic regurgitation can cause symptoms of heart failure, such as fatigue, shortness of breath and exercise intolerance.
Time Frame: 10 years post-implant
Population: Analysis population includes participants implanted with the Trifecta™ valve in 2007, 2008 and 2009 as part of the Trifecta™ IDE Study who consented to be enrolled in this study and who have aortic regurgitation assessment data available at 10 years post-implant.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 155
Participants
  None | 60
  Trivial | 53
  Mild | 30
  Moderate | 12
  Severe | 0

9. Other Pre Specified Outcome: Number of Participants by New York Heart Association (NYHA) Functional Class, Preoperatively and at 10 Years Post-Implant
Description: The New York Heart Association (NYHA) functional classification system relates heart failure symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Preoperative through 10 years
Population: Analysis population includes participants implanted with the Trifecta™ valve in 2007, 2008 and 2009 as part of the Trifecta™ IDE Study who consented to be enrolled in this study and have available Preoperative and/or 10-year NYHA classification data.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Previously Implanted With a Trifecta™ Valve
Number analyzed (Participants) | 329
Participants
  Preoperative: NYHA Class I | 23
  Preoperative: NYHA Class II | 166
  Preoperative: NYHA Class III | 133
  Preoperative: NYHA Class IV | 7
  10 Years: number analyzed (Participants) | 152
  10 Years: NYHA Class I | 111
  10 Years: NYHA Class II | 26
  10 Years: NYHA Class III | 14
  10 Years: NYHA Class IV | 1

ADVERSE EVENTS:
Time Frame: 10 Years
Description: Adverse event data collection includes all serious adverse events recorded in each participant from the time of their Trifecta™ implant under the Trifecta™ IDE study in 2007, 2008 and 2009 through the end of the Trifecta™ LTFU study in 2019. Non-serious adverse event data were not collected.
Groups:
- Subjects Previously Implanted With a Trifecta Valve: Subjects enrolled in this clinical study received the Trifecta valve during the investigational study that was conducted to obtain FDA approval. The Trifecta™ is a tri-leaflet stented pericardial valve designed for supra-annular placement in the aortic position.
Arm/Group | Subjects Previously Implanted With a Trifecta Valve
All-Cause Mortality (participants affected / at risk) | 67/329
Serious Adverse Events (participants affected / at risk) | 272/329
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Previously Implanted With a Trifecta Valve (N=329)
Anemia (Blood and lymphatic system disorders) | 8 (10)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Major Bleeding (Blood and lymphatic system disorders) | 42 (44)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrhythmias (Cardiac disorders) | 93 (122)
Endocarditis (Cardiac disorders) | 5 (5)
Heart Failure Signs and Symptoms (Cardiac disorders) | 34 (46)
Mitral Regurgitation (Cardiac disorders) | 4 (4)
Myocardial Ischemia (Cardiac disorders) | 26 (29)
Paravalvular Leak (Cardiac disorders) | 3 (3)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Structural Valve Deterioration, Explanted (Cardiac disorders) | 31 (31)
Structural Valve Deterioration, Transcatheter Valve-in-Valve Implant (Cardiac disorders) | 34 (34)
Structural Valve Deterioration without Reintervention (Cardiac disorders) | 19 (19)
Valve Thrombosis (Cardiac disorders) | 1 (1)
Diabetic Hyperglycemia (Endocrine disorders) | 1 (1)
Thyroid Disorders (Endocrine disorders) | 2 (3)
Eye Disorders (Eye disorders) | 4 (4)
Abdominal Hernias (Gastrointestinal disorders) | 7 (7)
Appendicitis (Gastrointestinal disorders) | 3 (5)
Esophageal Disorders (Gastrointestinal disorders) | 5 (5)
Vomiting, Diarrhea, Constipation (Gastrointestinal disorders) | 13 (16)
Intestinal Disorders (Gastrointestinal disorders) | 10 (12)
Death from Unknown Causes (General disorders) | 8 (8)
Dehydration (General disorders) | 3 (3)
Dizziness (General disorders) | 7 (7)
Fatigue (General disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Heat Stroke (General disorders) | 1 (1)
Hematoma (General disorders) | 4 (4)
Event Classification Unknown (General disorders) | 2 (2)
Biliary Obstruction (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 9 (10)
Bacteremia or Septicemia (Infections and infestations) | 5 (5)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 24 (31)
Wound Infections (Infections and infestations) | 20 (20)
Abdominal Abscess (Infections and infestations) | 2 (2)
Joint Disorders (Musculoskeletal and connective tissue disorders) | 55 (77)
Benign Lesions (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (33)
Delerium (Nervous system disorders) | 17 (17)
Siezure Disorders (Nervous system disorders) | 4 (5)
Concussion (Nervous system disorders) | 2 (2)
Psychiatric Disorders (Psychiatric disorders) | 2 (2)
Renal Disorders (Renal and urinary disorders) | 15 (16)
Urinary Tract Disorders (Renal and urinary disorders) | 24 (27)
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 7 (8)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 17 (19)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cellulitis (Skin and subcutaneous tissue disorders) | 6 (6)
Lacerations or Contusions (Skin and subcutaneous tissue disorders) | 3 (3)
Rashes, Eruptions And Exanthems (Skin and subcutaneous tissue disorders) | 2 (2)
Aortic Artery Disease (Vascular disorders) | 2 (2)
Carotid Artery Disease (Vascular disorders) | 4 (4)
Deep Vein Thrombosis (Vascular disorders) | 8 (9)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Disease (Vascular disorders) | 9 (13)
Thromboembolism (Vascular disorders) | 19 (21)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Air Embolism (Vascular disorders) | 1 (1)
Minor Bleeding (Blood and lymphatic system disorders) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 4 (4)
Foot Abscess (Infections and infestations) | 1 (1)
Klebsiella Infections (Infections and infestations) | 1 (1)
Fractures (Musculoskeletal and connective tissue disorders) | 8 (9)
Tendon, Ligament and Cartilage Disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Guillain-Barré Syndrome (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Respiratory Tract Signs and Symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Barotrauma (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT01593917/Prot_SAP_000.pdf